CLINICAL TRIAL: NCT05061056
Title: Neuromuscular Electrical Stimulation: Comparison of Carrier Frequencies, Bursts Durations and Duty Cycles in the Generation of Evoked Torque, Sensory Discomfort, Muscle Fatigue and Peripheral Oxygen Extraction
Brief Title: Effects of Neuromuscular Electrical Stimulation Parameters on Torque, Fatigue, and Oxygen Extraction
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Associate professor, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 47989121.6.0000.8093
Record Dates: First submitted 2021-09-09; First posted 2021-09-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Fatigue
Keywords: Healthy Young; Electric Stimulation Therapy; Evoked torque; Sensory discomfort; Peripheral oxygen extraction
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Russian current 10% (Experimental): Subjects will receive a interventions (Russian Current at 10% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Russian current 10%
- Russian current 20% (Experimental): Subjects will receive a interventions (Russian Current at 20% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Russian current 20%
- Aussie current 10% (Experimental): Subjects will receive a interventions (Aussie Current at 10% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Aussie current 10%
- Aussie current 20% (Experimental): Subjects will receive a interventions (Aussie Current at 20% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Aussie current 20%

INTERVENTIONS:
Other: Russian current 10% — Russian current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts
  Arms: Russian current 10%
Other: Russian current 20% — Russian current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 20% duty cycle - 4 ms bursts and 16 ms interbusrts
  Arms: Russian current 20%
Other: Aussie current 10% — Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts
  Arms: Aussie current 10%
Other: Aussie current 20% — Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 20% duty cycle - 4 ms bursts and 16 ms interbusrts
  Arms: Aussie current 20%

SUMMARY:
Neuromuscular Electrical Stimulation (NMES) can minimize muscle atrophy, complications related to muscle disuse and improved neuromuscular performance. However, it is still unclear the influence of specific physical parameters, including carrier frequency, burst duration, and duty cycle regarding the greater generation of evoked torque, sensory discomfort, muscle fatigue, and peripheral oxygen extraction. Thus, the aim of this study is to compare the effects of different NMES protocols applied to the triceps surae muscle for evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction in healthy individuals. This is a crossover, experimental, randomized, double-blind trial composed of apparently healthy participants. All NMES protocols will be tested on the same individual with randomization of the sequence of intervention protocols. There will be a total of 6 encounters with seven days between them. Session 1 will evaluate the anthropometric measures, the maximum intensity for each intervention protocol, and the sequence of intervention protocols for each individual will be randomized. Sessions 2, 3, 4, and 5 will be composed equally with the assessment of the maximum voluntary and evoked joint torque of the triceps surae muscle through the isokinetic dynamometer, evaluation of muscle fatigue through the H-reflex, M-wave, fatigue index, time-torque-integral, and recruitment curve, evaluation of peripheral oxygen extraction through NIRS (Near Infrared Spectroscopy), electromyographic signals to assessed the RMS (root mean square) and the median frequency, evaluation of the level of sensory discomfort through the Visual Analog Pain Scale and finally by the NMES protocol. The 6th session will be the replication of the 2nd session of each individual. The EENM protocols will be as follows: CR10% (Russian Current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts), CR20% (Russian Current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 20% of duty cycle - 4 ms bursts and 16 ms interbusrts), CA10% (Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 10% duty cycle - 2 ms of bursts and 18 ms interbusrts), CA20% (Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 20% of duty cycle - 4 ms of bursts and 16 ms interbusrts) all protocols will be performed on the triceps surae muscle.

DETAILED DESCRIPTION:
This is a crossover, experimental, randomized, double-blind trial composed of apparently healthy participants. The objective is to compare the effects of different NMES protocols applied to the triceps surae muscle for evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction. The effects of the types of neuromuscular electrical stimulation (NMES) protocols on the aforementioned outcomes will be evaluated in the same participant by randomizing the sequences of interventions for each visit in the laboratory. The study is considered double-blind, as individuals will not know the sequence of the protocols applied. The evaluator will also not know which protocol will be used at the time of the intervention. It will consist of a total of 6 sessions with seven days between them. In the first session, anthropometry, the maximum intensity level for each electrical stimulation protocol as well as the protocol sequence for each individual will be evaluated. From the second to the fifth session, the following will be considered: voluntary and evoked maximum joint torque of the triceps surae muscle, muscle fatigue through the evaluation of the H-reflex, M-wave, fatigue index, torque-time-integral and recruitment curve, peripheral oxygen extraction, electromyographic signals through RMS (root mean square) and median frequency, and level of sensory discomfort with the Visual Analog Scale (VAS). The last session will consist of the same electrical stimulation protocol from the second session of assessment. From the second to the fifth session will be composed by the following evaluation sequence: warm-up with six submaximal contractions with 6 seconds of duration and 10 seconds of rest between them; then the assessment of muscle fatigue; then three maximal isometric contractions, then three maximal evoked contractions; fatigue protocol at 20% of the maximum isometric contraction (this fatigue protocol will use the NMES sequence randomized in the first session, except on the fifth day that the NMES protocol used will be the same as the second day); after the fatigue protocol, three maximum evoked contractions will be performed again; then three maximal isometric contractions and at the end, the muscle fatigue evaluation will be performed again. The NMES protocols will be CR10% (Russian Current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts), CR20% (Russian Current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 20% of duty cycle - 4 ms of bursts and interbusrts of 16 ms), CA10% (Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts), CA20% (Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 20% duty cycle - 4 ms bursts and 16 interbusrts) ms) all protocols will be performed on the triceps surae muscle.

ELIGIBILITY:
Inclusion Criteria:

* Female and male, aged between 18-40 years,
* Be classified as physically active according to the International Physical Activity Questionnaire (IPAQ),
* The practice of just recreational physical activity,
* Achieve a minimum torque of 20% of the MVIC during the NMES
* Be at least three months without strength training

Exclusion Criteria:

* Present musculoskeletal dysfunction that may interfere with the tests, present intolerance to NMES in the triceps surae muscle,
* Use analgesics, antidepressants, tranquilizers, or other centrally acting agents
* Present cardiovascular or peripheral vascular problems, chronic diseases, neurological or muscle disorders that may impair the complete execution of the study design by the volunteer

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Submaximal voluntary isometric contraction of the triceps surae | 2 minutes
  Expressed in muscle strength, assessed using an isokinetic dynamometer
Maximum voluntary isometric contraction of the triceps surae | 5 minutes
  Expressed in muscle strength, assessed using an isokinetic dynamometer
Maximum evoked torque | 5 minutes
  Expressed by the description of muscle strength generated by electrical stimulation assessed by the isokinetic dynamometer
Torque evoked during the fatigue protocol | 20 minutes
  Expressed by the description of muscle strength generated by electrical stimulation assessed by the isokinetic dynamometer
Peripheral oxygen extraction | 40 minutes
  Expressed by peripheral oxygen consumption assessed by near-infrared spectroscopy from the beginning to the end of the sessions
Muscle fatigue assessment before the muscle fatigue protocol | 10 minutes
  Expressed by mechanical properties of plantar flexors and central activation relationship using the contraction interpolation technique
Assessment of muscle fatigue during the muscle fatigue protocol | 20 minutes
  Expressed by the muscle fatigue index through the decline in torque evoked from the beginning to the end of the protocol
Muscle fatigue assessment during the muscle fatigue protocol | 20 minutes
  Expressed by the decline in torque-time-integral from the beginning to the end of the protocol
Electromyographic signals | 40 minutes
  Expressed by the raw values of RMS and Median Frequency within a range of 500 ms throughout the entire session

SECONDARY OUTCOMES:
Sensory discomfort during maximum evoked torques | 10 seconds
  Measured through the Visual Analog Scale (1 - 10 cm) where 0 represents no discomfort and 10 represents greater discomfort
Sensory discomfort during fatigue protocol | 10 seconds
  Measured through the Visual Analog Scale (1 - 10 cm) where 0 represents no discomfort and 10 represents greater discomfort

CONTACTS AND LOCATIONS:
Overall Officials: João Durigan, PhD, Principal Investigator — University of Brasilia
Locations (1):
- João Luiz Q. Durigan, Brasília, Brasil, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baldi JC, Jackson RD, Moraille R, Mysiw WJ. Muscle atrophy is prevented in patients with acute spinal cord injury using functional electrical stimulation. Spinal Cord. 1998 Jul;36(7):463-9. doi: 10.1038/sj.sc.3100679. PMID 9670381
- [Result] Vaz MA, Baroni BM, Geremia JM, Lanferdini FJ, Mayer A, Arampatzis A, Herzog W. Neuromuscular electrical stimulation (NMES) reduces structural and functional losses of quadriceps muscle and improves health status in patients with knee osteoarthritis. J Orthop Res. 2013 Apr;31(4):511-6. doi: 10.1002/jor.22264. Epub 2012 Nov 8. PMID 23138532
- [Result] Delitto A, Strube MJ, Shulman AD, Minor SD. A study of discomfort with electrical stimulation. Phys Ther. 1992 Jun;72(6):410-21; discussion on 421-4. doi: 10.1093/ptj/72.6.410. PMID 1589461
- [Result] Dantas LO, Vieira A, Siqueira AL Jr, Salvini TF, Durigan JL. Comparison between the effects of 4 different electrical stimulation current waveforms on isometric knee extension torque and perceived discomfort in healthy women. Muscle Nerve. 2015 Jan;51(1):76-82. doi: 10.1002/mus.24280. PMID 24809656
- [Result] McLoda TA, Carmack JA. Optimal burst duration during a facilitated quadriceps femoris contraction. J Athl Train. 2000 Apr;35(2):145-50. PMID 16558623
- [Result] Liebano RE, Waszczuk S Jr, Correa JB. The effect of burst-duty-cycle parameters of medium-frequency alternating current on maximum electrically induced torque of the quadriceps femoris, discomfort, and tolerated current amplitude in professional soccer players. J Orthop Sports Phys Ther. 2013 Dec;43(12):920-6. doi: 10.2519/jospt.2013.4656. Epub 2013 Oct 30. PMID 24175604
- [Result] Vanderthommen M, Duteil S, Wary C, Raynaud JS, Leroy-Willig A, Crielaard JM, Carlier PG. A comparison of voluntary and electrically induced contractions by interleaved 1H- and 31P-NMRS in humans. J Appl Physiol (1985). 2003 Mar;94(3):1012-24. doi: 10.1152/japplphysiol.00887.2001. Epub 2002 Nov 27. PMID 12571132
- [Result] Paz IA, Rigo GT, Sgarioni A, Baroni BM, Frasson VB, Vaz MA. Alternating Current Is More Fatigable Than Pulsed Current in People Who Are Healthy: A Double-Blind, Randomized Crossover Trial. Phys Ther. 2021 Jun 1;101(6):pzab056. doi: 10.1093/ptj/pzab056. PMID 33561279
- [Result] Arpin DJ, Forrest G, Harkema SJ, Rejc E. Submaximal Marker for Investigating Peak Muscle Torque Using Neuromuscular Electrical Stimulation after Paralysis. J Neurotrauma. 2019 Mar 19;36(6):930-936. doi: 10.1089/neu.2018.5848. Epub 2018 Nov 16. PMID 30226407
- [Result] Botter A, Oprandi G, Lanfranco F, Allasia S, Maffiuletti NA, Minetto MA. Atlas of the muscle motor points for the lower limb: implications for electrical stimulation procedures and electrode positioning. Eur J Appl Physiol. 2011 Oct;111(10):2461-71. doi: 10.1007/s00421-011-2093-y. Epub 2011 Jul 28. PMID 21796408